CLINICAL TRIAL: NCT02068833
Title: Resolution of Microalbuminuria and Dysmetabolism Following Bariatric Surgery: Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: Johnson & Johnson (Industry); Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Sponsor
Other Study IDs: 20839
Record Dates: First submitted 2014-02-06; First posted 2014-02-21 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Microalbuminuria; Gastrectomy; Biliopancreatic Diversion With Duodenal Switch
Keywords: Microalbuminuria; Gastrectomy; Biliopancreatic Diversion With Duodenal Switch
MeSH Terms: interventions — Gastrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gastrectomy: Subjects in this group will undergo a gastrectomy only.
  Interventions: Procedure: Gastrectomy
- BPD-DS: Subjects in this group will undergo a BPD-DS surgery.
  Interventions: Procedure: BPD-DS

INTERVENTIONS:
Procedure: Gastrectomy
  Groups: Gastrectomy
Procedure: BPD-DS
  Groups: BPD-DS

SUMMARY:
Favorable effects of bariatric surgery have been demonstrated in particular regarding increased insulin sensitivity, decreased blood pressure, improved blood lipids and decreased cardiovascular risk. After surgery, weight loss also leads to improvement of the chronic inflammatory state related to obesity, a strong predictor of the metabolic status. Although obese patients are often affected with type 2 diabetes and hypertension, both related to renal impairment, the existence of a distinct mechanism by which obesity would cause chronic renal insufficiency has been suggested. The mechanisms underlying obesity-related nephropathy have been proposed to involve hyperfiltration, expansion of mesangial cells, hyperperfusion leading to proteinuria and glomerulosclerosis, as noted in obese dogs. In humans, improvements in renal function may be observed following bariatric surgery, although some reported a possibility of increased nephrolithiases. Whether biliopancreatic diversion and gastrectomy alone have similar effects is uncertain. More prospective studies are needed to assess the impact of all types of weight loss surgery to reverse chronic renal insufficiency.

The objective of this study is to document changes in microalbuminuria and metabolic parameters in patients with altered renal function undergoing bariatric surgery. Patients enrolled in the study will show renal function impairment as demonstrated by albumin/creatinine ratio alterations in 2 out of 3 measurements taking place before surgery. We will perform a prospective study of renal function markers (albumin/creatinine ratio) and metabolic parameters (blood lipids, glucose, insulin, inflammatory markers) before and 6, 12, 24 months after surgery in patients with microalbuminuria at study onset (albumin/creatinine ratio 2.0-20.0 mg/mmol in men and 2.8-28.0 mg/mmol in women). Data will be analysed with repeated measures analyses in both subgroup. Thereafter, a linear regression model will be created to adjust for potentially confounding factors such as hypertension and diabetes. We hypothesize that patients with severe obesity and altered renal function, whether they are diabetic or not, have improved microalbuminuria and metabolic parameters following biliopancreatic diversion with sleeve gastrectomy or sleeve gastrectomy alone. The extent of renal function recovery will correlate directly with metabolic improvements.

ELIGIBILITY:
Inclusion Criteria:

* Patient showing preoperative microalbuminuria (albumine/creatinine ratio between 2.0 and 20.0 in men and between 2.8 and 28.0 in women
* Men and Women between 18-60 years old;
* BMI ≥ 40 kg/m2 or between 35 and 40 kg/m2 if they have high-risk comorbidities;
* Subjects capable of understanding and being able to sign a consent form;
* Subjects capable of following the protocol directives, including the proposed visits (timeline);
* Subjects living within a reasonable distance from the hospital and capable of being present at all required visits.

Exclusion Criteria:

* Urinary infection;
* Hematuria (2+ or more) on 2 urinary analyses performed at 1 week interval;
* Hyperglycemia > 11 mmol/L at the time of the 2 urinary analyses;
* Known renal disease unrelated to hypertension or diabetes, normoalbuminuria, macroalbuminuria or proteinuria;
* Pregnant women or women who plan on becoming pregnant during the study, or women in fertile age range who refuse proper contraceptive methods during the study. (Must have negative pregnancy test at moment of enrolment and use medically acceptable contraception which include; oral contraceptives, injectable or implantable contraceptives, intrauterine devices or double-barrier method ie. condoms and diaphragm);
* Previous oesophagal, gastric or bariatric surgery;
* Irritable bowel syndrome, unexplained intermittent vomiting, severe abdominal pain, diarrhea or chronic constipation;
* History of duodenal or gastric ulcers;
* History of renal disease, hepatic disease (cirrhosis) or severe cardiac or pulmonary disease;
* Corticosteroid intake in the previous month;
* Presence of psychiatric problems or behavioral issues that could limit subject's capacity at understanding the procedure and to conform to medical/surgical recommendations;
* History of drug use or alcoholism in previous 12 months before study;
* History of inflammatory diseases of the gastro-intestinal tract (Esophagitis, varices, gastric or duodenal ulcers, Crohn's disease, congenital or acquired anomalies of the digestive tract).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will include patients 18 years and older with microalbuminuria (albumin/creatinine ratio between 2.0 and 20.0 mg/mmol in men and between 2.8 and 28.0 mg/mmol in women) planned to undergo either biliopancreatic diversion with sleeve gastrectomy or sleeve gastrectomy alone.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Changes in A/C Ratio | Baseline, 6, 12, 24 months
  * A/C Ratio
  * Weight Loss

CONTACTS AND LOCATIONS:
Locations (1):
- CRIUCPQ, Québec, Quebec, Canada